CLINICAL TRIAL: NCT04878679
Title: Effects of Combined Whole Body Electromiostimulation (WB-EMS) and Dynamic Movements on Motor and Cognitive Performance, Neurotrophic Factors and Alpha-synuclein in Parkinson's Disease
Brief Title: Effect of WB-EMS on Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Università degli studi di Roma Foro Italico (Other)
Collaborators: Giuseppe Calcagno (Unknown); Giovanni Fiorilli (Unknown); Andrea Buonsenso (Unknown); Marco Centorbi (Unknown)
Responsible Party: Principal Investigator, Alessandra di Cagno, Prof. Alessandra di Cagno, Università degli studi di Roma Foro Italico
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ForoItalico1
Record Dates: First submitted 2021-04-21; First posted 2021-05-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Strength training + WB-EMS" (Experimental): Strength training combined with WB-EMS : 2 times/week for 20 minutes
  Interventions: Other: Strenght training combined with WB-EMS
- Cardiovascular training + WB-EMS (Experimental): Cardiovascular training, using rowing machine, combined with WB-EMS : 2 times/week for 20 minutes
  Interventions: Other: Cardiovascular training with WB-EMS
- Control group (Active Comparator): No physical activity
  Interventions: Other: Control group

INTERVENTIONS:
Other: Strenght training combined with WB-EMS — Bodyweight exercise training combined with WB-EMS (2 times/week) with a 85Hz electrical impulse
  Arms: "Strength training + WB-EMS"
Other: Cardiovascular training with WB-EMS — Cardiovascular training , using the rowing machine, combined with WB-EMS (2 times/week) with a 7Hz electrical impulse
  Arms: Cardiovascular training + WB-EMS
Other: Control group — No physical activity
  Arms: Control group

SUMMARY:
The aim is to establish adequate and suitable protocols for PD patients and to determine the WB-EMS effects on muscle strength, balance, walking, cognitive functions,neurotrophic factors and alpha-synuclein. Thirty-six PD patients, aged from 50 to 80 years, will be recruited and randomly assigned to two experimental groups (EGs and EGc) and one control group (CG), in order to perform dynamic movements with WB-EMS. EGs will undergo to 12-20 minutes of progressive supervised WB-EMS (4 sec. 85 HZ and 4 sec. rests) combined to light dynamic movements, two-time per week for 12/24 weeks. EGe will undergo to 12-20 minutes of progressive supervised WB-EMS 7 Hz) combined with cardiovascular training with rowing machine. CG will not perform any type of physical activity. Pre and post intervention assessment will be carried out on the following areas: physical assessment, neurocognitive, neurotrophic factors and alpha-synuclein assesments. A 3 months follow-up will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age from 50 to 80 years old
* clinical diagnosis of parkinson's disease from 1 to 3 of Hoehn and Yahr Scale
* no partecipation to other physical activity program

Exclusion Criteria:

* MMSE values < 24
* inability to walk 6 minutes without assistance
* use of medications and other things that may affect cognitive and motor functions
* presence of contraindications in the use of WB-EMS

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
REPETITIONS NUMBER CHANGE | 14 Weeks
  30S ARM CURL TEST
REPETITIONS NUMBER CHANGE | 14 Weeks
  30S SIT TO STAND TEST;
TIME(S) CHANGE | 14 Weeks
  SODA POP TEST ;
TIME(S) CHANGE | 14 Weeks
  8 FEET UP AND GO TEST ;
DISTANCE (M) CHANGE | 14 Weeks
  6 MINUTE WALKING TEST
UPPER LIMB STRENGHT CHANGE | 14 Weeks
  HAND GRIP TEST
LOWER BODY FLEXIBILITY | 14 Weeks
  CHAIR SIT AND REACH TEST
BALANCE AND STABILITY TEST CHANGE | 14 Weeks
  TINETTI BALANCE AND GAIT EVALUATION TEST
NUMBER OF ERRORS CHANGE | 14 Weeks
  STROOP TEST;
NUMBER OF ERRORS CHANGE | 14 Weeks
  REY AUDITORY VERBAL LEARNING TEST
TIME(S) CHANGE | 14 Weeks
  STROOP TEST
TIME(S) CHANGE | 14 Weeks
  TRAIL MAKING TEST CHANGE
NEUROTROPHIC FACTORS CHANGE | 14 Weeks
  BLOOD DRAW
ALPHA-SYNUCLEIN CHANGE | 14 Weeks
  BLOOD DRAW

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra di Cagno, Principal Investigator — Università degli studi di Roma Foro Italico
Locations (1):
- Università degli Studi del Molise, Campobasso, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] di Cagno A, Buonsenso A, Centorbi M, Manni L, Di Costanzo A, Casazza G, Parisi A, Guerra G, Calcagno G, Iuliano E, Soligo M, Fiorilli G; WB-EMS Parkinson's Group. Whole body-electromyostimulation effects on serum biomarkers, physical performances and fatigue in Parkinson's patients: A randomized controlled trial. Front Aging Neurosci. 2023 Feb 9;15:1086487. doi: 10.3389/fnagi.2023.1086487. eCollection 2023. PMID 36845654
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886